CLINICAL TRIAL: NCT02042378
Title: A Phase 2, Open-Label Study of Rucaparib in Patients With Pancreatic Cancer and a Known Deleterious BRCA Mutation
Brief Title: A Study of Rucaparib in Patients With Pancreatic Cancer and a Known Deleterious BRCA Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: pharmaand GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-338-023
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma
Keywords: BRCA; BRCA mutation; germline BRCA; somatic BRCA; PARP inhibitor; rucaparib; CO-338; PF 01367338; AG 14699; Clovis; Clovis Oncology; RucaPanc
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rucaparib (Experimental): All patients will take oral tablets twice daily with 8 oz (240 mL) of water on an empty stomach or with food; 28-day cycles of treatment. Doses should be taken as close to 12 hours apart as possible, preferably at the same times every day. Tablets should be swallowed whole.
  Interventions: Drug: Rucaparib

INTERVENTIONS:
Drug: Rucaparib — All patients will take oral tablets twice daily with 8 oz (240 mL) of water on an empty stomach or with food; 28-day cycles of treatment. Doses should be taken as close to 12 hours apart as possible, preferably at the same times every day. Tablets should be swallowed whole.
  Other Names: CO-338; PF 01367338; AG 14699

SUMMARY:
The purpose of this study is to determine whether oral rucaparib is effective in the treatment of patients with locally advanced or metastatic pancreatic cancer and a known deleterious BRCA mutation.

DETAILED DESCRIPTION:
Rucaparib is an orally available, small molecule inhibitor of poly-adenosine diphosphate [ADP] ribose polymerase (PARP) that inhibits a specific DNA repair pathway known as base excision repair (BER). PARP inhibitors (PARPi) have been shown to effectively kill tumors with a defect in BRCA1 or BRCA2. Clinical benefit has been observed in patients with a gBRCA mutation as well as in those with a somatic BRCA (sBRCA) mutation. Clinical data have also shown that pancreatic cancer patients with a gBRCA mutation benefit from PARPi treatment. Clinical activity of PARP inhibitors in BRCA-mutated pancreatic cancer combined with the paucity of 2nd line therapies support evaluation of rucaparib in pancreatic cancer patients known to harbor a deleterious BRCA mutation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of pancreatic cancer (ductal adenocarcinoma and related subtypes eligible; endocrine and neuroendocrine tumors excluded)
* Received at least 1, but no more than 2, chemotherapy-based regimens for locally advanced or metastatic disease and has relapsed or progressive disease. Patients no longer able to continue treatment with chemotherapy due to intolerable toxicity may be considered for study participation provided that radiology assessment confirms either stable disease or disease progression (i.e. no response to treatment)
* Documented deleterious or suspected deleterious (or equivalent interpretation) BRCA mutation (germline or somatic) as assessed by a local laboratory
* Measurable disease

Exclusion Criteria:

* Presence of another active cancer
* Prior treatment with any PARP inhibitor, including rucaparib. Patients treated with prior iniparib are eligible.
* Symptomatic and/or untreated central nervous system metastases.
* Clinical evidence of malabsorption and/or any other gastrointestinal disorder or defect that would, in the opinion of the investigator, interfere with the absorption of rucaparib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) per RECIST v1.1 as assessed by the investigator | Screening, within 7 days prior to the start of every 3rd cycle of treatment, and Treatment Discontinuation Visit. Study to last for ~3 years.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) per RECIST v1.1 as assessed by independent radiology review | Screening, within 7 days prior to the start of every 3rd cycle of treatment, and Treatment Discontinuation Visit. Study to last for ~3 years.
Duration of Response (DOR) by RECIST v1.1 | Screening, within 7 days prior to the start of every 3rd cycle of treatment, and Treatment Discontinuation Visit. Study to last for ~3 years.
PFS defined as the occurrence of disease progression according to RECIST v1.1, as assessed by the investigator, or death from any cause | Screening, within 7 days prior to the start of every 3rd cycle of treatment, and Treatment Discontinuation Visit. Study to last for ~3 years.
Overall Survival (OS) | To be performed continually from first dose of study drug through discontinuation, then every 4 weeks until death, loss to follow-up, withdrawal of consent from study, or closure of the study. Study to last for ~3 years.
Incidence of adverse events (AEs), clinical laboratory abnormalities, and dose modifications | Continuously from signing of informed consent to 28 days after the last dose. Study to last for ~3 years.
Trough (Cmin) level rucaparib concentrations | Cycle 1 Day 15, Cycle 2 Day 15, Cycle 3 Day 1, and Cycle 4 Day 1. Study to last for ~3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Giordano, Study Director — Clovis Oncology, Inc.
Locations (8):
- United States (5):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mayo Clinic, Rochester, Minnesota
  - New York University, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Israel (3):
  - Rambam Healthcare Campus, Haifa
  - Hadassah Hebrew University Hospital (Sharett Institute of Oncology), Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv